CLINICAL TRIAL: NCT05485831
Title: Observational, Prospective, Multicenter Study of Epidyolex® (Cannabidiol CBD 100 mg/ml) Oral Solution, as Adjunctive Treatment for Seizures Associated With Lennox- Gastaut Syndrome (LGS), Dravet Syndrome (DS) and Tuberous Sclerosis Complex (TSC)
Brief Title: Epidyolex® in Lennox Gastaut, Dravet Syndrome and Tuberous Sclerosis Complex: an Observational Study in ITALY
Acronym: EpiTALY
Status: Recruiting | Type: Observational
Sponsor: Jazz Pharmaceuticals (Industry)
Collaborators: Advice Pharma Group srl (Industry)
Responsible Party: Sponsor
Other Study IDs: JZP926-525
Record Dates: First submitted 2022-07-29; First posted 2022-08-03 (Actual); Last update posted 2025-12-31 (Actual); Status verified 2025-12

CONDITIONS: Lennox Gastaut Syndrome; Dravet Syndrome; Tuberous Sclerosis Complex
Keywords: seizures; Epidyolex; cannabidiol oral solution
MeSH Terms: conditions — Lennox Gastaut Syndrome; Epilepsies, Myoclonic; Tuberous Sclerosis; Seizures | interventions — Cannabidiol; Solutions

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Lennox Gastaut, Dravet Syndrome, and Tuberous Sclerosis Complex: Participants ≥2 years of age diagnosed with LGS, DS, and TSC.
  Interventions: Drug: Epidiolex 100 mg/mL Oral Solution

INTERVENTIONS:
Drug: Epidiolex 100 mg/mL Oral Solution — As prescribed in routine clinical practice in Italy.

SUMMARY:
This is a prospective, observational study on approximately 70-100 Real World participants affected by LGS, DS, or TSC treated with Epidyolex® as prescribed in the summary of product characteristics. The eligible participants are expected to participate in the study for a duration of 52 weeks of treatment.

DETAILED DESCRIPTION:
This observational study evaluates a Real-World population of children and adult participants affected by LGS, DS, and TSC and the effect of therapy with Epidyolex® administered according to clinical practice on epileptic symptoms. The study will assess specific scales, questionnaires, and the satisfaction of the caregivers and the participants/tutors.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients, and minor patients ≥ 2 years old diagnosed with LGS, DS or TSC.
* Clinical decision, taken by the physician, to initiate Epidyolex®
* Adult participants, parents or legal representatives must be willing and able to give informed consent/assent for participation in the study.

Exclusion Criteria:

* Participants currently using or have used recreational, medicinal cannabis, or cannabinoid-based products within the three months prior to study entry and are unwilling to abstain from these products for the duration of the study.
* Any reason, according to Investigator's judgment, able to compromise compliance with procedures outlined in the study There will not be any other specific exclusion criteria; however, contraindications, special warnings, and precautions for use as detailed in the Summary of Product Characteristics (SmPC) (particularly related to raising of aspartate aminotransferase [AST], alanine aminotransferase [ALT], and total bilirubin) will have to be considered by the treating physician.

Min Age: 2 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: The study will comprise of 70-100 male and female participants, aged ≥ 2 years, diagnosed with LGS, DS, and TSC. The decision to prescribe Epidyolex® as adjunctive therapy for seizures associated with LGS, DS, and TSC will be entirely independent of including the participant in the study.
Sampling Method: Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2025-02-24 (Actual); Primary Completion 2026-01 (Estimated); Study Completion 2026-01 (Estimated)

PRIMARY OUTCOMES:
Number of Participants Remaining on Therapy from Enrollment | Baseline up to Week 52 post-dose.
  Treatment retention will be evaluated through the proportion of participants remaining on therapy from the enrollment visit (baseline, V0) to each study visit (Weeks 4 [V1], 16 [V2], 28 [V3], 40 [V4], 52 [V5]).

SECONDARY OUTCOMES:
Average Number of Seizure-Free Days in the Last 28 Days | Weeks 4 (V1), 16 (V2), 28 (V3), 40 (V4) and 52 (V5)
Longest Duration of Seizure Free Days in the Last 28 Days | Weeks 4 (V1), 16 (V2), 28 (V3), 40 (V4) and 52 (V5)
Average Maintenance Dose of Epidyolex® | Weeks 4 (V1), 16 (V2), 28 (V3), 40 (V4) and 52 (V5)
Maximum Maintenance Dose of Epidyolex® | Weeks 4 (V1), 16 (V2), 28 (V3), 40 (V4) and 52 (V5)
Type, Dosage, and Frequency of Concomitant Anti-Seizure Medications (ASMs) | Weeks 4 (V1), 16 (V2), 28 (V3), 40 (V4) and 52 (V5)
Number of Participants Reducing Number/Dosage of Concomitant Medication Related to Epilepsy | Weeks 4 (V1), 16 (V2), 28 (V3), 40 (V4) and 52 (V5)
Change from Baseline to Week 28 (V3) in the Child Behavior Check List (CBCL) | Baseline to week 28 (V3) post-dose.
  The CBCL is a standardized form that parents fill out to describe their children's behavioral and emotional problems(e.g., anxiety, depression, social problems). The CBCL is also scored on (optional) competence scales for activities, social relations, school and total competence. The CBCL consists of 113 questions, scored on a three-point Likert scale (0=absent, 1= occurs sometimes, 2=occurs often). A higher score indicates a worse outcome.
Change from Baseline to Week 52 (V5) in the Child Behavior Check List (CBCL) | Baseline to week 52 (V5) post-dose.
  The CBCL is a standardized form that parents fill out to describe their children's behavioral and emotional problems(e.g., anxiety, depression, social problems). The CBCL is also scored on (optional) competence scales for activities, social relations, school and total competence. The CBCL consists of 113 questions, scored on a three-point Likert scale (0=absent, 1= occurs sometimes, 2=occurs often). A higher score indicates a worse outcome.
Change from Baseline to Week 28 (V3) in the Visual Analog Scale (VAS) of 10 Non-seizure Related Outcomes (NSRO) | Baseline to week 28 (V3) post-dose.
  VAS assessments are based on 10 NSRO (i.e., Alertness, Sleep Disorder, Motor Skills, Attention, Cognition, Communication, Behavior, Emotional/Social Functioning, Activities of Daily Living, and Participation). VAS is measured on a scale of 0-100; a score of 0 indicates a better outcome, and a score of 100 indicates a worse outcome.
Change from Baseline to Week 52 (V5) in the VAS of 10 NSRO | Baseline to week 52 (V5) post-dose.
  VAS assessments are based on 10 NSRO (i.e., Alertness, Sleep Disorder, Motor Skills, Attention, Cognition, Communication, Behavior, Emotional/Social Functioning, Activities of Daily Living, and Participation). VAS is measured on a scale of 0-100; a score of 0 indicates a better outcome, and a score of 100 indicates a worse outcome.
Average Caregiver Global Impression of Change (CGIC) Score at Week 28 (V3) | Week 28 (V3) post-dose.
  The CGIC evaluates efficacy and quality of life. At enrollment the investigator will be asked to write a brief description of the patient's overall condition as a memory aid for assessment at each subsequent appointment. The CGIC comprises of the following question: "Since your child started treatment, please assess the status of your child's overall condition (comparing their condition now to their condition before treatment) using the scale below." The questionnaire is rated on a seven-point scale: "Very Much Improved" (1); "Much Improved" (2);Slightly Improved" (3); "No Change" (4); "Slightly Worse" (5); "Much Worse" (6); "Very Much Worse" (7). A score of 1 indicates a better outcome and a score of 7 indicates a worse outcome.
Average CGIC Score at Week 52 (V5) | Week 52 (V5) post-dose.
  The CGIC evaluates efficacy and quality of life. At enrollment the investigator will be asked to write a brief description of the patient's overall condition as a memory aid for assessment at each subsequent appointment. The CGIC comprises of the following question: "Since your child started treatment, please assess the status of your child's overall condition (comparing their condition now to their condition before treatment) using the scale below." The questionnaire is rated on a seven-point scale: "Very Much Improved" (1); "Much Improved" (2);Slightly Improved" (3); "No Change" (4); "Slightly Worse" (5); "Much Worse" (6); "Very Much Worse" (7). A score of 1 indicates a better outcome and a score of 7 indicates a worse outcome.
Average Caregiver Global Impression of Change in Seizure Duration (CGICSD) Score at Week 28 (V3) | Week 28 (V3) post-dose.
  The CGICSD comprises the following question to be rated on a three-point scale for each seizure subtype: Since the patient started treatment, please assess the average duration of the patient's seizures (comparing their condition now to their condition before treatment) using the scale below. The scale markers are: 1=Average duration of seizures has decreased; 2=Average duration of seizures has stayed the same; 3=Average duration of seizures has increased. Higher scores indicate a worse outcome.
Average CGICSD Score at Week 52 (V5) | Week 52 (V5) post-dose.
  The CGICSD comprises the following question to be rated on a three-point scale for each seizure subtype: Since the patient started treatment, please assess the average duration of the patient's seizures (comparing their condition now to their condition before treatment) using the scale below. The scale markers are: 1=Average duration of seizures has decreased; 2=Average duration of seizures has stayed the same; 3=Average duration of seizures has increased. Higher scores indicate a worse outcome.
Average Physician Global Impression of Change (PGIC) Score at Week 28 (V3) | Week 28 (V3) post-dose.
  The PGIC evaluates efficacy and quality of life. At enrollment the investigator will be asked to write a brief description of the patient's overall condition as a memory aid for assessment at each subsequent appointment. The PGIC comprises of the following question: "Please assess the change in the patient's general functional abilities since enrolment." The questionnaire is rated on a seven-point scale: "Very Much Improved" (1); "Much Improved" (2);Slightly Improved" (3); "No Change" (4); "Slightly Worse" (5); "Much Worse" (6); "Very Much Worse" (7). A score of 1 indicates a better outcome and a score of 7 indicates a worse outcome.
Average PGIC Score at Week 52 (V5) | Week 52 (V5) post-dose.
  The PGIC evaluates efficacy and quality of life. At enrollment the investigator will be asked to write a brief description of the patient's overall condition as a memory aid for assessment at each subsequent appointment. The PGIC comprises of the following question: "Please assess the change in the patient's general functional abilities since enrolment." The questionnaire is rated on a seven-point scale: "Very Much Improved" (1); "Much Improved" (2);Slightly Improved" (3); "No Change" (4); "Slightly Worse" (5); "Much Worse" (6); "Very Much Worse" (7). A score of 1 indicates a better outcome and a score of 7 indicates a worse outcome.

CONTACTS AND LOCATIONS:
Locations (18):
- Italy (18):
  - Policlinico Sant'Orsola di Bologna, Bologna
  - NPI AOU Mater Domini Università Magna Graecia, Catanzaro
  - Università degli studi "G. D'annunzio" Chieti, Chieti
  - Azienda Ospedaliera Universitaria Meyer Neurologia Pediatrica, Florence
  - Istituto Gaslini Neurologia Pediatrica e Malattie Muscolari, Genova
  - AOU Gaetano Martino, Messina
  - Centro Regionale Epilessia - ASST Santi Paolo e Carlo, Milan
  - ASST Grande Ospedale metropolitano Niguarda, Milan
  - Azienda Ospedaliera Universitaria Federico II, Napoli
  - AOU Maggiore della Carità di Novara, Novara
  - AOU di Padova, Padua
  - Policlinico Tor Vergata, Roma
  - IRCCS Ospedale Pediatrico Bambin Gesù, Roma
  - Fondazione Policlinico Universitario Agostino Gemelli - IRCCS-NPI, Roma
  - Azienda Ospedaliero Universitaria Sant'Andrea, Roma
  - Ospedale Casa del sollievo e della sofferenza, San Giovanni Rotondo
  - AOU Città della Salute PO Molinette, Torino
  - Azienda Ospedaliero Universitaria delle Marche, Torrette

IPD SHARING:
Plan to Share IPD: No